CLINICAL TRIAL: NCT02352857
Title: Postprandial Glycaemic and Insulinaemic Responses After Consumption of Minicakes Containing FOS in Adults
Brief Title: Glycaemic and Insulinaemic Responses After Consumption of FOS.
Acronym: GLYCOFOS-cake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: Syral (Industry)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, MD, Endocrinologist, Nutritionist, Institut Pasteur de Lille
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2013-A00785-40
Record Dates: First submitted 2013-11-25; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Glycaemia
Keywords: Fructo-oligosaccharides; Sugar-reduced foods; Postprandial glucose response
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar (Placebo Comparator): Control group consuming sponge cakes containing in total 24g of dextrose.
  Interventions: Other: Sugar
- FOS (Experimental): Group consuming sponge cakes in which 30% of the dextrose was replaced by FOS.
  Interventions: Other: FOS

INTERVENTIONS:
Other: Sugar — 100g of sponge cakes made with 24g of dextrose.
  Arms: Sugar
Other: FOS — 100g of sponge cakes made with 19.4g of dextrose and 9.1g of FOS.
  Arms: FOS

SUMMARY:
The study aims to evaluate the glycaemic and insulinaemic response of short-chain fructo-oligosaccharides (scFOS) used to replace sugars (e.g. dextrose) in foods.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 25.0 kg/m² (included);
* Ready to keep the same volume of physical activity and the same dietary habits during the study and particularly 24 hours before each visit;
* Be used to have breakfast;
* Non-smoker for at least 3 months;
* For the female participant: not being pregnant or breastfeeding and using efficient birth control;
* Signed the consent form;
* Able to follow the instructions of the study;
* Health insured;
* Accepted to be included in the National Registry for biomedical research Volunteers (Fichier VRB, Volontaires Recherches Biomédicales).

Exclusion Criteria:

* Fasting blood glucose over 6.1 mmol/L (1.10 g/L) (or diabetes treated or not);
* Fasting blood cholesterol over 6.35 mmol/L;
* Fasting blood triglycerides over 1.70 mmol/L (or history of insulinoma);
* Fasting blood insulin under 20 mU/L;
* Fasting HbA1c under 7%;
* History of hypercholesterolemia, hypertension, diabetes or glucose intolerance treated or not;
* History of dietary allergies or coeliac disease;
* History of digestive system disease susceptible to modify digestion or absorption like Crohn's disease;
* Somatic or psychiatric disorders;
* Renal insufficiency (kidney failure);
* SGOT or ALAT over 52.5 U/L;
* Smoker;
* Consuming more than 3 alcoholic beverage a day;
* Weight varied 3 kg the last 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Glycaemic response | 2 hours and 5 minutes
  Blood glucose kinetics with 7 points. Analysis of the Area under the curve of glucose.

SECONDARY OUTCOMES:
Insulinaemic response | 2 hours and 5 minutes
  Blood insulin kinetics with 7 points. Analysis of the Area under the curve of insulin.
Blood glucose peak (Cmax) | One-time data (the highest one) within the 2hrs 5mins kinetics.
  Peak of blood glucose during kinetics.
Blood insulin peak (Cmax) | One-time data (the highest one) within the 2hrs 5mins kinetics.
  Peak of blood insulin during kinetics.
Glucose Tmax : time to reach the peak of blood glucose | One time within the 2hrs 5mins kinetics.
Insulin Tmax : time to reach the peak of blood insulin | One time within the 2hrs 5mins kinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel LECERF, MD, Principal Investigator — Institut Pasteur de Lille
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France